CLINICAL TRIAL: NCT04528238
Title: Multicentric, Randomized, Open-label Study to Assess the Impact of Relaxing Visual Immersion (RVI) on Reducing Anxiety During Intravenous Cancer Treatment in Cancer Patients.
Brief Title: Impact of Relaxing Visual Immersion on Anxiety During Anti-cancer Treatment.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: following the covid health crisis the study has not begun
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMAVANX
Record Dates: First submitted 2020-07-29; First posted 2020-08-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxing Visual Immersion (Experimental): The patients will benefit a Relaxing Visual Immersion during the intravenous treatment for their cancer.
  Interventions: Other: Relaxing Visual Immersion
- No sensitive stimulation (No Intervention): The patients will not receive Relaxing Visual Immersion during the intravenous treatment for their cancer.

INTERVENTIONS:
Other: Relaxing Visual Immersion — During the intravenous treatment for cancer, a nature movie will be projected on the ceiling of the room, along with natural sounds or a relaxing music. The patient will choose the movie or movies he wants to watch and can decide to stop the Relaxing Visual Immersion (RVI) at any time. The RVI is a system that does not isolate the patient from his familiar or medical entourage and which integrates virtual scenarios in the environment of care.
  Arms: Relaxing Visual Immersion

SUMMARY:
Since the 60's and 70's, the soar of audiovisual technologies allowed the development of virtual reality (VR). These technologies were then adapted to help reducing anxiety and pain during medical procedures. For visual or audio stimulation, the use of glasses or helmet is frequent. However, little is know about the efficacy of technologies which are not isolating the patient from his real environment during medical care. With this study, the investigators will assess the impact of this kind of sensitive stimulation without isolating the patient, on reducing the anxiety during intravenous treatment in patients with cancer. The machine the investigators are using is projecting relaxing nature movies on the ceiling of the room, with nature sounds or relaxing music.

DETAILED DESCRIPTION:
The diagnosis of cancer and the treatments used may be the cause, for the patient, of a significant emotional and psychological anxiety. For many years, several studies have evaluated the impact of visual and sensitive techniques on the well-being of the patient: landscaping of gardens,use of positive distraction means (decoration, brightness of spaces, photographs, layout of natural scenes, aquarium installation, etc.). The objective of these studies was to give to the patient a contact with nature reinforcing the positive emotions and reducing stress.

A randomized study including 37 patients who will undergo flexible sigmoidoscopy of diagnosis, to receive during the intervention, audio stimulation, audio and visual stimulation by glasses (Virtual IO, 1000 Leonora), or no stimulation. Audio and visual stimulation reduced abdominal discomfort (measured using visual analog scale VAS) and a decrease in anxiety (measured by the Stress Symptom Ratings scale) compared to the group without stimulation (p <0.05), but without solid evidence given the small number of patients with an imprecise randomization.

Other distraction systems using paintings of nature scenes combined with a listening to the sounds of nature were used during bronchoscopy: 80 patients were randomized (distraction systems versus control group without stimulation): the decrease in pain (rated on a 5-point scale from poor to excellent) was significantly greater in the intervention versus control group (p <0.015). There was no significant effect on anxiety measured by the S-STAI scale compared to the control group (with a 6 point difference between groups). Another Chinese prospective randomized controlled trial (Lee et al. 2004), conducted on 165 patients, has shown that visual and audio distraction (by Eyetrek system, Olympus) could reduce the need for sedatives used during colonoscopy compared to the group with visual distraction only and in the distraction-free control group (p <0.01). From the years 1960-1970, the development of digital audiovisual technologies allowed to develop virtual reality techniques. The term "virtual reality" (VR) refers to a computer technology that simulates artificially the user's environment, with which the user can interact. In oncology, virtual reality (VR) techniques have been used in 3 situations :

- during painful procedures: A randomized controlled study conducted on 30 adolescents with cancer who will undergo a lumbar puncture, analyzed the impact of VR glasses on pain assessed by VAS and the feedback of the patients. There was no statistically significant difference between 2 groups but pain scores were lower in the VR group (The mean VAS in the VR group was 7 points with a range ranging from 0 to 48 while in the control group the average was 9 points with a range from 0 to 59).

Another randomized study conducted on 59 children with cancer whose treatments required access to a subcutaneous venous device assessed the value of VR distraction, non-virtual distraction and the absence of distraction. Reductions in pain and anxiety have been observed (measured by VAS) in children using VR distraction but were not significant given the small sample size. However the reduction of the heart rate was significant in the VR distraction group (p <0.05).

- during hospitalization: This situation is considered stressful because it is linked to a change in the state of health and because it introduces stressful conditions like lack of autonomy, privacy, etc.

A study showed on 19 hospitalized patients with metastatic cancer, exposed to 4 sessions of 30 minutes for 1 week with a VR headset, an increase in joy over the 4 sessions (before and after the test, p <0.009) and a decrease in sadness over the 2nd session (before and after the test, p <0.003).

Another study showed on 33 hospitalized patients with metastatic cancer under the same conditions as the Banos study, an increase in positive emotions and a decrease in negative emotions after each session (p <0.05).

- during the chemotherapy infusion to reduce the symptoms related to the treatment or disease: A study evaluated the interest of VR by head-mounted display (Sony PC Glasstron PLM-S700) in 16 women aged 50 years and older during chemotherapy infusions. The symptoms such as anxiety and fatigue were assessed (STAI scale and revised Piper scale PFS). Patients were randomized to 2 chemotherapy sessions with the use of VR head-mounted display for one session and without stimulation for the other session. A decrease in anxiety immediately after the session was shown in this small number of patients (p = 0.10). On the other hand, there was no difference for fatigue but the study was carried out only on one session of RV.

It was showed a benefit of VR in 123 patients with breast, lung or colon cancer, receiving 2 chemotherapy sessions: participants were randomized according to a cross-over design in order to receive the VR intervention (by i-Glasses SVGA HeadMounted Display helmet) during one chemotherapy session and to receive during the other session no VR intervention (control arm), each patient being their own control. This technique was using a laptop, VR headset, and software. The Symptom Distress Scale was used to assess symptoms of distress immediately after the session and 48 hours after the session. No significant difference was found for the symptoms of distress between the session receiving the VR intervention and the session not receiving the intervention of VR. However, the study only assessed the use of VR over a single treatment session. The patients who received the VR technique had a decrease in anxiety during the initial session of chemotherapy (decrease of 3.34 points, p = 0.01). In addition, the perception of the time during the chemotherapy session was significantly altered, making the session more tolerable because it is shorter and thus validating the distraction capacity of this intervention.

When it comes to physical variables (vital signs), 4 studies found a significant difference in heart rate with a lower rate in the Virtual Reality group.

However, few studies in oncology have looked at non-isolating devices for VR (without helmet or glasses), therefore without excluding the patient from his environment. This non-isolating technology has also been considered as being able to offer the patient a more secure environment.

The purpose of this study is to assess the impact of this kind of stimulation during the intravenous treatment in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over.
* Patient with cancer (any location) who need to receive an intravenous (IV) cancer treatment (adjuvant, neoadjuvant or palliative) when taking initial disease burden or upon relapse (the IV treatments concomitant with radiotherapy are also possible).
* Patients scheduled for at least 3 consecutive sessions of IV anti-cancer treatment.
* Patient under health insurance plan.
* Information and signature of informed consent by the patient to participate in the study.

Exclusion Criteria:

* Pregnant women.
* Vulnerable patient (psychiatric illness, detainee, under legal protection, emancipated child).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of RVI on anxiety during the first intravenous cancer treatment session in cancer patients treated or not by anxiolytics | Baseline : first visit for intravenous anti-cancer treatment.
  Assessment of anxiety using the State-Trait Anxiety Inventory (STAI). The difference in the STAI-State anxiety score (STAI form Y-A) between e and after intervention will be studied in each group. A difference of at least 5 points of the change average before and after intervention between the experimental group and the control group will be considered as the minimum clinically significant difference.

SECONDARY OUTCOMES:
Assessment of pain felt. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using a visual analog scale.
Assessment of asthenia. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using the Piper's Revised Fatigue Scale.
Assessment of nausea. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using a visual analog scale.
Assessment of psychological distress. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using the Distress Thermometer Scale.
Assessment of the perception of elapsed time. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using a specific questionnaire designed for this study.
Assessment of the quality of patient - caregiver communication. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using a specific questionnaire designed for this study, for the caregiver point of view.
Assessment of the vital signs. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Taking blood pressure before and after each treatment session.
Assessment of the vital signs. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Taking cardiac rate before and after each treatment session.
Assessment of the undesirable effects linked to the RVI. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Collection of the adverse events (drought eye, headache, dizziness).
Assessment of the anxiety. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using the State-Trait Anxiety Inventory (STAI).
Analysis of the taking anti-anxiety treatments during anti-cancer treatment session | Up to 2 years, during 3 anti-cancer treatment sessions.
  Harvesting prescribed doses of anxiolytics during anti-cancer treatment sessions.
Assessment of the quality of life. | Up to 2 years, during 3 anti-cancer treatment sessions.
  Using the QLQ-C30 questionnaire.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berto R. The role of nature in coping with psycho-physiological stress: a literature review on restorativeness. Behav Sci (Basel). 2014 Oct 21;4(4):394-409. doi: 10.3390/bs4040394. PMID 25431444
- [Background] Schweitzer M, Gilpin L, Frampton S. Healing spaces: elements of environmental design that make an impact on health. J Altern Complement Med. 2004;10 Suppl 1:S71-83. doi: 10.1089/1075553042245953. PMID 15630824
- [Background] Lembo T, Fitzgerald L, Matin K, Woo K, Mayer EA, Naliboff BD. Audio and visual stimulation reduces patient discomfort during screening flexible sigmoidoscopy. Am J Gastroenterol. 1998 Jul;93(7):1113-6. doi: 10.1111/j.1572-0241.1998.00339.x. PMID 9672340
- [Background] Drahota A, Ward D, Mackenzie H, Stores R, Higgins B, Gal D, Dean TP. Sensory environment on health-related outcomes of hospital patients. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD005315. doi: 10.1002/14651858.CD005315.pub2. PMID 22419308
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899
- [Background] Lee DW, Chan AC, Wong SK, Fung TM, Li AC, Chan SK, Mui LM, Ng EK, Chung SC. Can visual distraction decrease the dose of patient-controlled sedation required during colonoscopy? A prospective randomized controlled trial. Endoscopy. 2004 Mar;36(3):197-201. doi: 10.1055/s-2004-814247. PMID 14986215
- [Background] Chirico A, Lucidi F, De Laurentiis M, Milanese C, Napoli A, Giordano A. Virtual Reality in Health System: Beyond Entertainment. A Mini-Review on the Efficacy of VR During Cancer Treatment. J Cell Physiol. 2016 Feb;231(2):275-87. doi: 10.1002/jcp.25117. PMID 26238976
- [Background] Sander Wint S, Eshelman D, Steele J, Guzzetta CE. Effects of distraction using virtual reality glasses during lumbar punctures in adolescents with cancer. Oncol Nurs Forum. 2002 Jan-Feb;29(1):E8-E15. doi: 10.1188/02.ONF.E8-E15. PMID 11845217
- [Background] Gershon J, Zimand E, Pickering M, Rothbaum BO, Hodges L. A pilot and feasibility study of virtual reality as a distraction for children with cancer. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1243-9. doi: 10.1097/01.chi.0000135621.23145.05. PMID 15381891
- [Background] Banos RM, Espinoza M, Garcia-Palacios A, Cervera JM, Esquerdo G, Barrajon E, Botella C. A positive psychological intervention using virtual reality for patients with advanced cancer in a hospital setting: a pilot study to assess feasibility. Support Care Cancer. 2013 Jan;21(1):263-70. doi: 10.1007/s00520-012-1520-x. Epub 2012 Jun 13. PMID 22688373
- [Background] Espinoza M, Banos RM, Garcia-Palacios A, Cervera JM, Esquerdo G, Barrajon E, Botella C. Promotion of emotional wellbeing in oncology inpatients using VR. Stud Health Technol Inform. 2012;181:53-7. PMID 22954828
- [Background] Schneider SM, Ellis M, Coombs WT, Shonkwiler EL, Folsom LC. Virtual reality intervention for older women with breast cancer. Cyberpsychol Behav. 2003 Jun;6(3):301-7. doi: 10.1089/109493103322011605. PMID 12855087
- [Background] Schneider SM, Hood LE. Virtual reality: a distraction intervention for chemotherapy. Oncol Nurs Forum. 2007 Jan;34(1):39-46. doi: 10.1188/07.ONF.39-46. PMID 17562631
- [Background] Schneider SM, Kisby CK, Flint EP. Effect of virtual reality on time perception in patients receiving chemotherapy. Support Care Cancer. 2011 Apr;19(4):555-64. doi: 10.1007/s00520-010-0852-7. Epub 2010 Mar 26. PMID 20336327
- [Background] Gershon J, Zimand E, Lemos R, Rothbaum BO, Hodges L. Use of virtual reality as a distractor for painful procedures in a patient with pediatric cancer: a case study. Cyberpsychol Behav. 2003 Dec;6(6):657-61. doi: 10.1089/109493103322725450. PMID 14756933
- [Background] Klosky JL, Tyc VL, Srivastava DK, Tong X, Kronenberg M, Booker ZJ, de Armendi AJ, Merchant TE. Brief report: Evaluation of an interactive intervention designed to reduce pediatric distress during radiation therapy procedures. J Pediatr Psychol. 2004 Dec;29(8):621-6. doi: 10.1093/jpepsy/jsh064. PMID 15491984